CLINICAL TRIAL: NCT02913729
Title: Pre- Versus Postoperative Accelerated Partial Breast Irradiation in Early Stage Breast Cancer Patients
Brief Title: Pre- Versus Postoperative Accelerated Partial Breast Irradiation
Acronym: PAPBI-2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15PAP; NL53862.031.15 (Other: CCMO)
Record Dates: First submitted 2016-02-04; First posted 2016-09-26 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer; Cancer of the Breast; Neoplasms, Breast
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- radiotherapy in arm 1 (Experimental): pre-operative accelerated partial breast irradiation
  Interventions: Radiation: partial breast irradiation
- radiotherapy in arm 2 (Active Comparator): post-operative accelerated partial breast irradiation
  Interventions: Radiation: partial breast irradiation

INTERVENTIONS:
Radiation: partial breast irradiation — irradiation
  Other Names: partial breast radiotherapy; accelerated breast irradiation

SUMMARY:
Most of the local recurrences (LR) found after breast-conserving therapy are within or close to the tumor bed. This pattern of recurrence was confirmed by studies of breast conserving surgery without adjuvant irradiation and by the update of the NSABP B-06 trial. In the EORTC boost trial, however, 29% of all LR were found outside the area of the original tumor. Still, a recent review of Breast Conserving Therapy (BCT) trials showed that the site of local recurrences after BCT was mostly in the tumor bed, with less than 10% of LR elsewhere in the breast. This led to the concept of partial breast irradiation. With accelerated partial breast irradiation (APBI), a limited volume of breast tissue is irradiated, allowing for a higher dose per fraction compared to whole breast irradiation (WBI), which is favorable considering the low alpha/beta ratio, and thus higher sensitivity to high dose per fraction.

DETAILED DESCRIPTION:
Patients will undergo a partial accelerated breast irradiation pre-or postoperative of 5 x 5.2 Gy

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 51 years
* clinical stage tumor-1-2 (≤ 3 cm)
* cN0
* Grade I or grade II (biopsy)
* Histologically proven invasive ductal adenocarcinoma
* Unifocal lesions on mammogram and MRI (small satellite lesions adjacent to the tumor are accepted as long as it is suitable for local excision to be determined by the participating centre)
* World Health Organization performance status ≤ 2
* Life expectancy ≥ 5 years
* Written informed consent

Exclusion Criteria:

* Distant metastases
* Lobular invasive carcinomas
* Pure Ductal Carcinoma in situ (DCIS) without invasive tumor
* Grade III in biopsy
* Triple negative tumors
* HER2neu positive tumors
* Lymphvascular invasion in biopsy
* TNM pathologic stage N1-3
* pN+ (micro- or macrometastases)
* Multicentric / multifocal disease on mammogram or MRI
* Diffuse calcifications on mammogram (Birads 3, 4 or 5)
* Prior treatment for the protocol tumor (no surgery, no neoadjuvant chemotherapy or neoadjuvant hormonal therapy, no previous radiotherapy)
* Previous contralateral breast cancer
* Other neoplasms in the last 5 years with the exception of:
* Basal cell carcinoma of the skin
* Adequately treated carcinoma in situ of the cervix
* Planned oncoplastic resection with tissue displacement
* No social security affiliation/health insurance
* Participation in another clinical trial that interferes with the locoregional treatment of this protocol
* It is expected that dosimetric constraints cannot be met, ie, lung/heart constraints or if the ratio PTV/ipsilateral breast >30%

Min Age: 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Cosmetic outcome | 3 years
  cosmetic effect will be measured by comparing the treated breast with the contralateral breast. Cosmetic effect will be scored in three different ways: by digital photographs, patient's questionnaires and specialist's questionnaires. These data will result in an overall cosmetic outcome, scored as excellent, good, fair or poor.

SECONDARY OUTCOMES:
tumor response | 6 weeks
  pathologic response will be measured in the removed tissue
postoperative complications | 6 weeks
  The expected acute surgical complication rate is approximately 16%. A stopping rule is set at 15% for complications that require hospitalization (including intravenous antibiotics) and re-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Scholten, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (6):
- France (2):
  - Institut Curie, Saint-Cloud
  - Institut Gustave-Roussy, Villejuif
- Netherlands (2):
  - Antoni van Leeuwenhoek, Amsterdam
  - University Medical Center Utrecht (UMCU), Utrecht
- Champilamaud Cancer Center, Lisbon, Portugal
- University General Hospital Valencia-Erasa, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
data from this clinical trial will be shared with the previous PAPBI clinical trial

REFERENCES:
- [Background] Bartelink H, Horiot JC, Poortmans PM, Struikmans H, Van den Bogaert W, Fourquet A, Jager JJ, Hoogenraad WJ, Oei SB, Warlam-Rodenhuis CC, Pierart M, Collette L. Impact of a higher radiation dose on local control and survival in breast-conserving therapy of early breast cancer: 10-year results of the randomized boost versus no boost EORTC 22881-10882 trial. J Clin Oncol. 2007 Aug 1;25(22):3259-65. doi: 10.1200/JCO.2007.11.4991. Epub 2007 Jun 18. PMID 17577015
- [Background] Cajucom CC, Tsangaris TN, Nemoto T, Driscoll D, Penetrante RB, Holyoke ED. Results of salvage mastectomy for local recurrence after breast-conserving surgery without radiation therapy. Cancer. 1993 Mar 1;71(5):1774-9. doi: 10.1002/1097-0142(19930301)71:53.0.co;2-v. PMID 8448741
- [Background] Elkhuizen PH, van de Vijver MJ, Hermans J, Zonderland HM, van de Velde CJ, Leer JW. Local recurrence after breast-conserving therapy for invasive breast cancer: high incidence in young patients and association with poor survival. Int J Radiat Oncol Biol Phys. 1998 Mar 1;40(4):859-67. doi: 10.1016/s0360-3016(97)00917-6. PMID 9531371
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Osborne MP, Borgen PI, Wong GY, Rosen PP, McCormick B. Salvage mastectomy for local and regional recurrence after breast-conserving operation and radiation therapy. Surg Gynecol Obstet. 1992 Mar;174(3):189-94. PMID 1542833
- [Background] Sanders ME, Scroggins T, Ampil FL, Li BD. Accelerated partial breast irradiation in early-stage breast cancer. J Clin Oncol. 2007 Mar 10;25(8):996-1002. doi: 10.1200/JCO.2006.09.7436. PMID 17350949
- [Background] Veronesi U, Volterrani F, Luini A, Saccozzi R, Del Vecchio M, Zucali R, Galimberti V, Rasponi A, Di Re E, Squicciarini P, et al. Quadrantectomy versus lumpectomy for small size breast cancer. Eur J Cancer. 1990;26(6):671-3. doi: 10.1016/0277-5379(90)90114-9. PMID 2144153